CLINICAL TRIAL: NCT02467309
Title: Association of Serum 25-hydroxyvitamin D Levels and Outcomes in Children With Bacterial Meningitis
Brief Title: Vitamin d Levels in Children With Bacterial Meningitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gang Liu (Other)
Responsible Party: Sponsor-Investigator, Gang Liu, director, chief physician, professor, Beijing Children's Hospital
Organization: Beijing Children's Hospital (Other)
Other Study IDs: 20150203
Record Dates: First submitted 2015-03-18; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Bacterial Meningitis
MeSH Terms: conditions — Meningitis, Bacterial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether deficiency of Vitamin D has association with outcomes of children with bacterial meningitis.

DETAILED DESCRIPTION:
Vitamin D deficiency has been proved in serious diseases patients, including patients in shock, however, few study have been done about association between deficiency of Vitamin D and outcomes of children with bacterial meningitis.

in our study, we will observe incidence of complication and severity of complication between patients who have different Vitamin D status.

ELIGIBILITY:
Inclusion Criteria:

* Probable bacterial meningitis patients: Clinical manifestation (Any person with sudden onset of fever (> 38.5 °C rectal or 38.0 °C axillary) and one of the following signs: neck stiffness, altered consciousness or other meningeal sign) with cerebrospinal fluid examination showing at least one of the following:

A. turbid appearance; B.leukocytosis (> 100 cells/mm3); C.leukocytosis (10-100 cells/ mm3) AND either an elevated protein (> 100 mg/dl) or decreased glucose (< 40 mg/dl)

* Confirmed bacterial meningitis patients: A case that is laboratory-confirmed by growing (i.e. culturing) or identifying (i.e. by Gram stain or antigen detection methods) a bacterial pathogen (Hib, pneumococcus or meningococcus) in the cerebrospinal fluid or from the blood in a child with a clinical syndrome consistent with bacterial meningitis

Exclusion Criteria:

* Congenital immunodeficiency patients
* HIV patients
* Patients with corticosteroid treatment for long time
* Patients with disorders in adrenal gland and pituitary gland and hypothalamus
* Patients with tuberculosis

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients who are diagnosed with bacterial meningitis in infectious diseases department of Beijing Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
vitamin d level change | change in serum vitamin d level from baseline to 28 days after initial hospitalization
  Serum vitamin d level will be detected in the first day of hospitalization and twenty-eighth day of hospitalization, no vitamin d supplementation during this time

SECONDARY OUTCOMES:
Clinical assessment of disease severity with Glasgow score | 1 day
  Disease severity will be assessed with Glasgow score in the first day of hospitalization
Clinical assessment of disease severity with Glasgow score | 7 day
  Disease severity will be assessed with Glasgow score in the seventh day of hospitalization
Clinical assessment of disease severity with Glasgow score | 28 day
  Disease severity will be assessed with Glasgow score in the twenty-eighth day of hospitalization
Clinical assessment of disease severity with pediatric critical illness score | 1 day
  Disease severity will be assessed with pediatric critical illness score in the first day of hospitalization
Clinical assessment of disease severity with pediatric critical illness score | 7 day
  Disease severity will be assessed with pediatric critical illness score in the seventh day of hospitalization
Clinical assessment of disease severity with pediatric critical illness score | 28 day
  Disease severity will be assessed with pediatric critical illness score in the twenty-eighth day of hospitalization
Clinical assessment of disease severity with cerebrospinal fluid examination | 1 day
  Cerebrospinal fluid examination including white blood cell count, protein concentration and glucose concentration in cerebrospinal fluid
Clinical assessment of disease severity with cerebrospinal fluid examination | 7 day
  Cerebrospinal fluid examination including white blood cell count, protein concentration and glucose concentration in cerebrospinal fluid
Clinical assessment of disease severity with cerebrospinal fluid examination | 28 day
  Cerebrospinal fluid examination including white blood cell count, protein concentration and glucose concentration in cerebrospinal fluid
Assessment of complications | 1 day
  Assessment of complications include whether patients have complications, which kind of complication patients suffered, and whether needing surgical therapy.
Assessment of complications | 7 day
  Assessment of complications include whether patients have complications, which kind of complication patients suffered, and whether needing surgical therapy.
Assessment of complications | 28 day
  Assessment of complications include whether patients have complications, which kind of complication patients suffered, and whether needing surgical therapy.